CLINICAL TRIAL: NCT02518165
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Trial to Assess the Effects of A Proprietary Spearmint Extract on Cognitive Performance, Mood, and Sleep in Men and Women
Brief Title: The Effects of A Proprietary Spearmint Extract on Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kemin Foods LC (Industry)
Collaborators: MusclePharm Sports Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 14HUS003
Record Dates: First submitted 2015-07-30; First posted 2015-08-07 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Mood; Cognitive Performance; Sleep
Keywords: Cognitive Domain: Speed; Cognitive Domain: Reaction Time; Cognitive Domain: Attention; Cognitive Domain: Executive Function; Cognitive Domain Memory; Sleep Quality; Sleep Efficiency
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proprietary spearmint extract (Active Comparator): Subjects randomized into the active treatment group will be asked to consume 900 mg/day of the proprietary spearmint extract.
  Interventions: Dietary Supplement: Proprietary spearmint extract
- Microcrystalline cellulose (Placebo Comparator): Subjects randomized into the placebo group will be asked to consume 900 mg/day of the excipient, microcrystalline cellulose.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Proprietary spearmint extract — Water extracted spearmint extract
  Arms: Proprietary spearmint extract
Other: Placebo — Microcrystalline Cellulose
  Arms: Microcrystalline cellulose

SUMMARY:
This study was designed to evaluate the chronic effects of a proprietary spearmint extract over 90 days of supplementation on aspects of cognitive performance (cognitive function and active reaction time), subjective mood, and sleep quality in healthy men and women.

ELIGIBILITY:
Inclusion Criteria:

* Men and pre-menopausal women, 18-50 years of age.
* Body mass index 18.5-29.99 kg/m2, inclusive or body mass index 30.0-34.99 kg/m2 and body fat via bioimpedance <39% for women aged 18-39y, <40% for women aged 40-50y, <25% for men aged 18-39y, <28% for men aged 40-50y.
* Participant has at least a high school diploma or the equivalent.
* Participant is recreationally active.
* Participant is judged by the Investigator to be in general good health.
* Participant understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigators.

Exclusion Criteria:

* Participant is unable to understand and/or perform required tests.
* Participant is unwilling to maintain normal dietary (including vitamins and supplements), exercise, sleep and medication patterns throughout the study.
* Participant is a habitual consumer of mint tea defined as >8oz per day.
* Participant is regularly taking a cognitive enhancing supplement.
* Participant has a history or presence of a clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorder.
* Participant has a sleep disorder or occupation where sleep during the overnight hours is irregular.
* Participant is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
* Participant is a current user of tobacco (defined as tobacco use within the previous 6 months).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Choice reaction time as assessed by the Makoto Arena Device | Change from baseline after 90 days of supplementation

SECONDARY OUTCOMES:
Cognitive function (speed, reaction time, attention, executive function, memory, and motor speed) as assessed by a computerized test battery | Change from baseline after 90 days of supplementation
Subjective mood as assessed using a Likert scale questionnaire | Change from baseline after 90 days of supplementation
Subjective sleep quality and efficiency as assessed using Likert and visual analog scale questionnaires | Change from baseline after 90 days of supplementation or between group comparisons at day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan R Moon, PhD, Principal Investigator — MusclePharm Sports Science Institute
Locations (1):
- Musclepharm Sports Science Institute, Denver, Colorado, United States

REFERENCES:
- [Derived] Falcone PH, Tribby AC, Vogel RM, Joy JM, Moon JR, Slayton CA, Henigman MM, Lasrado JA, Lewis BJ, Fonseca BA, Nieman KM, Herrlinger KA. Efficacy of a nootropic spearmint extract on reactive agility: a randomized, double-blind, placebo-controlled, parallel trial. J Int Soc Sports Nutr. 2018 Dec 12;15(1):58. doi: 10.1186/s12970-018-0264-5. PMID 30541572